CLINICAL TRIAL: NCT02896868
Title: A Multiple-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3041658 in Patients With Skin Diseases
Brief Title: A Study of LY3041658 in Participants With Skin Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 15165; I7P-MC-DSAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05-01

CONDITIONS: Skin Diseases; Psoriasis
MeSH Terms: conditions — Skin Diseases; Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY3041658 (Experimental): LY3041658 administered intravenously (IV) once every two weeks over 6 weeks (four doses).
  Interventions: Drug: LY3041658
- Placebo (Placebo Comparator): Placebo administered IV once every two weeks over 6 weeks (four doses).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3041658 — Administered IV.
  Arms: LY3041658
Drug: Placebo — Administered IV.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the safety and tolerability of the study drug known as LY3041658 in participants with certain types of skin diseases. The study will measure how the body absorbs, breaks down and gets rid of LY3041658. It will last about 127 days for each participant, not including screening. This study is for research purposes only, and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Investigator confirmed diagnosis of certain skin diseases for at least 6 months.
* Active skin lesions that are not responding to standard therapies.
* Willing to undergo pre- and post-treatment skin biopsies of lesions.

Exclusion Criteria:

- Have other skin diseases that may interfere with evaluation of the specified skin disease being studied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11-08 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Dosing Day 1 through Day 127

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3041658 | Dosing Day 1 through Day 127
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) During Dosing Interval at Steady State (AUCss) of LY3041658 | Dosing Day 1 through Day 127
Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of LY3041658 | Dosing Day 1 through Day 127

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Parexel Early Phase Unit at Glendale, Glendale, California
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - PAREXEL-Phase 1 Baltimore Harbor Hospital Center, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

REFERENCES:
- See also: Click here for more information about this study: A Study of LY3041658 in Participants With Skin Diseases — https://www.lillytrialguide.com/en-US/studies/skin-disease/DSAB#?postal=